CLINICAL TRIAL: NCT00204399
Title: Examining Physician Counseling to Promote Adoption of Physical Activity: A Controlled Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: HSF2001
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2000-05

CONDITIONS: No Specific Conditions Are Being Examined

INTERVENTIONS:
Behavioral: Telephone counseling support

SUMMARY:
The purpose of this study is to systematically test the efficacy of two physician-based interventions in changing physical activity patterns of adults over a 20-month period.

DETAILED DESCRIPTION:
Although physicians typically counsel for other risk factors of CVD, they are less likely to counsel for increasing levels of physical activity. This is surprising for two reasons: First, physical activity has been identified as an independent modifiable risk factor for CVD. Second, there is a high prevalence of physical inactivity among Canadians. The purpose of the current study is to examine interventions that are designed to promote adoption and maintenance of physical activity through physician recommendations and counseling. The primary outcome measures include possible differences in levels of self-reported physical activity. In addition, several behavioral predictors typically associated with physical activity will be assessed (e.g., self-efficacy, social support, anticipated benefits & enjoyment, and barriers). There are several unique aspects to this research including: 1) the fact that it compares two types of delivery systems 2) the examination of physical activity patterns over an extended period of time has not been done previously with this type of intervention, and as such, also forms another unique feature of this proposal 3) physician intervention for physical activity has not been done in Canada previously. If the intervention is found effective, the program will add significant value to health services in Saskatchewan and Canada. For instance, the program will enhance the role of physicians in promoting physical activity without increasing the cost of health-care delivery, and with a minimal investment of time required by the physician and his/her staff.

Comparison: To assess the efficacy of the interventions, a quasi experimental design will compare an intervention with a standard control condition. All physicians will be trained to use a standardized protocol to deliver PACE exercise counseling to sedentary patients during one office visit. In the intervention condition, patients will be randomly assigned to receive reminder calls from a research assistant who will provide suggestions as to possible physical activity resources in the community that could be used.

ELIGIBILITY:
Inclusion Criteria:

* ambulatory adults

Exclusion Criteria:

* cardiovascular disease
* respiratory disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2001-07; Study Completion 2004-12

PRIMARY OUTCOMES:
The primary outcome measures include possible differences in levels of self-reported physical activity.

SECONDARY OUTCOMES:
In addition, several behavioral predictors typically associated with physical activity will be assessed (e.g., self-efficacy, social support, anticipated benefits & enjoyment, and barriers).

CONTACTS AND LOCATIONS:
Overall Officials: Kevin S Spink, Ph.D., Principal Investigator — University of Saskatchewan